CLINICAL TRIAL: NCT05452330
Title: Comparison of the Effectiveness of Connective Tissue Massage and Classical Massage in Patients With Migraine
Brief Title: The Effect of Two Different Massages on Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Begum Kara Kaya, Clinical investigator, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Migren
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-07

CONDITIONS: Headache, Migraine; Manuel Therapy
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Connective tissue massage
  Interventions: Other: Connective tissue massage
- Group 2 (Experimental): Classical massage
  Interventions: Other: Classical massage

INTERVENTIONS:
Other: Connective tissue massage — Connective tissue massage will be applied with short and long pulling strokes to create a reflex effect for 2 days a week, a total of 8 weeks.
  Arms: Group 1
Other: Classical massage — Classical massage will be applied with the techniques of stroking, kneading, and friction for 2 days a week, a total of 8 weeks.
  Arms: Group 2

SUMMARY:
The study aims to compare the effects of connective tissue massage on pain severity, attack frequency and duration, migraine-related disability, and quality of life in patients diagnosed with migraine, by comparing them with the classical massage.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers with a migraine diagnosis
* Taking only analgesics for migraine treatment and continuing their routines
* No problem in reading, writing and understanding Turkish

Exclusion Criteria:

* Having any other neurological problems
* Who had been injected with botulinum toxin in the last 3 months

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 8 weeks
  The intensity of pain perceived by the subjects will be evaluated with a valid method, the Visual Analogue Scale (VAS). The higher numbers show higher pain intensities.

SECONDARY OUTCOMES:
Migraine Related Disability | 8 weeks
  The Migraine Disability Assessment Scale (MIDAS), which is considered valid and reliable, will be used to evaluate the migraine-related disability. The higher scores indicate an increase in the severity of the disability.
The Quality of Life | 8 weeks
  The patients' quality of life will be evaluated with the 24-hours Quality of Life in Migraine Scale (24-Hr-MQoLQ), which is valid and reliable. The increase in the score obtained from the scale indicates an increase in the quality of life.
Perceived Patient-Reported Change | 8th week (one week)
  The change perceived by the patients after the intervention will be evaluated with the Global Rating of Change Scale (GROC). According to the scale, it is expressed as "-2: I am much worse, -1: I am worse, 0: No change, 1: I am better, 2: I am much better".
The general descriptive demographic information | 8 weeks
  The general descriptive demographic information of the participants such as age and gender; migraine family history, duration of the complaints, attack frequency and duration will be questioned with a form prepared by the researchers.

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Özdinçler, PhD, Study Chair — Biruni University
Locations (1):
- Biruni University, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No